CLINICAL TRIAL: NCT02389205
Title: Rehabilitation Department of Tri-Service General Hospital
Brief Title: The Effect of Functional Activities and Balance Ability With Taping in Subjects of Hemophilia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Chan Yuan-Chi, physical therapist, Tri-Service General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: TSGH-105-165
Record Dates: First submitted 2014-11-04; First posted 2015-03-17 (Estimated); Last update posted 2015-03-19 (Estimated); Status verified 2015-03

CONDITIONS: Hemophilia
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- control group (Placebo Comparator): physical therapy
- kinesio group (Active Comparator): kinesio taping for ankle joint
  Interventions: Other: kinesio group

INTERVENTIONS:
Other: kinesio group — kinesio group, The kinesio Taping® Method is a definitive rehabilitative taping technique that is designed to facilitate the body's natural healing process while providing support and stability to muscles and joints without restricting the body's range of motion as well as providing extended soft tissue manipulation to prolong the benefits of manual therapy administered within the clinical setting.
  The effect of intervention may affected by the varying durations and frequencies of exercise, different state of arthropathy and joint range of motion limitations of ankle , etc.
  Arms: kinesio group

SUMMARY:
Background Hemophilia is a sex-linked genetic disorders. When the joint or the muscles is bleeding, it may cause haemarthrosis, synovium, cartilage tissue thickening, joint activity (Range of Motion) decreasing and other musculoskeletal and related disorder. Patients will produce pain in the action, compensatory action occurs, thus causing recurrent of bleeding, and joint damage. There is high rate of ankle joint bleeding in hemophilia. The ankle articular joint disease will affect lower limbs activities, and the functional activities will impaired.

Review studies, in addition to physical therapy, Kinesio taping is a common intervention to improve other subjects' static balance, proprioception, functional ankle stability, correct poor posture.

The main intervention of this study is physical therapy and Kinesio taping, expect to improve the stability and muscular strength of lower extremities, and balance, correcting gait and lower extremity functional activities of subjects with hemophilia.

DETAILED DESCRIPTION:
Methods:

This study is a randomized controlled trial, the subjects were randomly divided into two groups, the control group received physical therapy once a week for a period of three months; experimental group received the same physical therapy in addition to treatment, but each will be accepted Kinesio taping. Experiments group carried out before and after the relevant tests, including: muscle strength, balance, lower extremity functional activities. The participants will be followed for the duration of physical therapy , an expected average of 3 months.

ELIGIBILITY:
Inclusion Criteria:

* subject of Hemophilia
* 20-65 years old

Exclusion Criteria:

* Any history of surgery

Ages: 20 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-04; Primary Completion 2015-11 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
standing balance ability (biodex balance system) | 3 months
  biodex balance system

CONTACTS AND LOCATIONS:
Overall Officials: Chen Liang-Cheng, Study Director — Director of Rehabilitation department

REFERENCES:
- [Result] Rodriguez-Merchan EC. Orthopaedic problems about the ankle in hemophilia. J Foot Ankle Surg. 2012 Nov-Dec;51(6):772-6. doi: 10.1053/j.jfas.2012.06.005. Epub 2012 Jul 10. PMID 22785085